CLINICAL TRIAL: NCT02444143
Title: A Pharmacokinetic Analysis of Tacrolimus ER Dosing in Obese Kidney Transplant Recipients
Acronym: Tacrolimus ER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia West-Thielke, Director of Clinical Research, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-XXXX
Record Dates: First submitted 2014-11-20; First posted 2015-05-14 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Immunosuppression; Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBW (Active Comparator): tacrolimus extended release 0.15 mg/kg/day based on Ideal Body Weight (IBW)
  Interventions: Drug: tacrolimus extended release
- ABW (Experimental): tacrolimus extended release 0.15 mg/kg/day based on adjusted Body Weight (aBW)
  Interventions: Drug: tacrolimus extended release

INTERVENTIONS:
Drug: tacrolimus extended release
  Other Names: Astagraf XL

SUMMARY:
Tacrolimus extended release (Astagraf) has recently been approved by the FDA as a once a day dosing regimen. This formulation has the potential to improve compliance. Current dosing recommendation for the extended release formulation in renal transplant is 0.15 mg/kg/day administered once daily in the morning. There are no specifications on appropriate dosing in obese patients or on whether to use actual, ideal or and adjusted weight. It will be advantageous to understand the pharmacokinetics of this medication in the obese to determine the appropriate dosing regimen. In this study, obese patients will be randomized to receive tacrolimus extended release 0.15 mg/kg/day based on either ideal body weight (IBW) or adjusted body weight (aBW).

DETAILED DESCRIPTION:
Tacrolimus exhibits significant inter- and intra-individual variability of its absorption and metabolism. Because of this variability, standard dosing is not an accurate predictor of drug exposure. In clinical use, tacrolimus whole blood trough concentrations are measured to ensure efficacy and safety. Furthermore, the relatively low bioavailability of tacrolimus is thought to be a result of the combination of poor water-solubility, pre-systemic metabolism of tacrolimus in the gastrointestinal tract and activity of the P-glycoprotein efflux pump found in the enterocytes of the GI tract. Tacrolimus is extensively metabolized by the cytochrome P-450 system (CYP3A). The plasma protein binding of tacrolimus is approximately 99%. Tacrolimus is bound mainly to albumin and alpha-1-acid glycoprotein. The distribution of tacrolimus between blood and plasma depends on several factors including hematocrit, temperature at the time of plasma separation, drug concentration, and plasma protein concentration.

Pharmacodynamic studies have revealed that, depending on time following transplantation, maintaining whole blood trough levels between 5 and 20 ng/mL provides adequate protection against acute rejection and limits the occurrence of adverse events. The management of tacrolimus blood levels is complicated by variable intra- and inter-patient absorption, interaction with food and concomitant medications, and the relatively low bioavailability of tacrolimus from the Prograf formulation (17 ± 10% in adult kidney transplant patients).

Previous studies examining immunosuppressants have shown that drug levels in the immediate post-transplant period are a major determinant of subsequent acute cellular rejection. It is known that tacrolimus (TAC) < 10 ng/mL is associated with increased rates of acute cellular rejection by one month post-transplant.

There is controversy regarding the appropriate dosing weight to use for immunosuppressants (IS). Weights use range from ideal body weight (IBW) to total body weight (TBW) depending on the institution and drug being dosed. This becomes particularly important in the obese population when there are significant differences between IBW and TBW. Our institution has always used IBW for the dosing of all IS due to concerns for nephrotoxicity with initial high blood levels of tacrolimus. The concern in obese patients is that the investigators are underdosing this population that could be at higher risk for rejection due to higher circulating concentrations of pro-inflammatory cytokines. The introduction of the novel use of a robotic transplantation procedure at our institution for this patient population has led to increasing numbers of transplant in obese recipients; therefore, the investigators decided to re-evaluate our dosing protocol. Data from an internal study at UIC show that our use of IBW for tacrolimus dosing is not sufficient for the obese population (body mass index [BMI] ≥30). The dose used through month 3 was closer to 0.1 mg/kg/day when total body weight was utilized. However, the use of an adjusted body weight (aBW) is common for medication dosing in obese patients. Adjusted body weight is calculated if the TBW is greater than 30% of the calculated IBW. aBW = IBW + 0.4(TBW - IBW). There is limited data available supporting the use of either IBW or aBW in dosing tacrolimus within obese patients as these patients are typically excluded from most clinical trials, particularly the pharmacokinetic trials. In addition, no literature is available comparing the two dosing weights to determine which leads to therapeutic concentrations most effectively.

Summary and Present Study Tacrolimus extended release (Astagraf) has recently been approved by the FDA as a once a day dosing regimen. This formulation has the potential to improve compliance. Current dosing recommendation for the extended release formulation in renal transplant is 0.15 mg/kg/day administered once daily in the morning. There are no specifications on appropriate dosing in obese patients or on whether to use actual, ideal or and adjusted weight. It will be advantageous to understand the pharmacokinetics of this medication in the obese to determine the appropriate dosing regimen. In this study, obese patients will be randomized to receive tacrolimus extended release 0.15 mg/kg/day based on either ideal body weight (IBW) or adjusted body weight (aBW).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a recipient of a living donor or deceased donor kidney only transplant
2. Subject is > 18 years of age
3. BMI≥30 on POD 0

Exclusion Criteria:

1. Multi-organ transplant
2. Subjects taking tacrolimus pre-transplant (i.e. positive crossmatch transplants or re-transplants)
3. Patients undergoing simultaneous sleeve gastrectomy at the time of transplant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02-28 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Hospital & Health Sciences System, Chicago, Illinois, United States

REFERENCES:
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Jasiak-Panek NM, Wenzler E, Patel S, Thielke JJ, Progar K, Patel S, Brandt S, Huang YJ, Benedetti E, West-Thielke PM. A randomized, open-label pharmacokinetic trial of tacrolimus extended-release dosing in obese de novo kidney transplant recipients. Clin Transplant. 2019 Aug;33(8):e13640. doi: 10.1111/ctr.13640. Epub 2019 Jul 1. PMID 31206808

RESULTS

PARTICIPANT FLOW:
Groups:
- Ideal Body Weight- Tacrolimus Extended Release: tacrolimus extended release (Astagraf) 0.15 mg/kg/day based on Ideal Body Weight (IBW)
- Adjusted Body Weight-Tacrolimus Extended Release: tacrolimus extended release (Astagraf) 0.15 mg/kg/day based on adjusted Body Weight (aBW)
Period: Overall Study
Arm/Group | Ideal Body Weight- Tacrolimus Extended Release | Adjusted Body Weight-Tacrolimus Extended Release
Started | 10 | 10
Completed | 10 | 9 (1 patient withdrawal)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ideal Body Weight- Tacrolimus Extended Release | Adjusted Body Weight-Tacrolimus Extended Release | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.6) | 47.7 (14.3) | 54 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Body Mass Index greater than or equal to 30 on Post Operative Day 0 [Count of Participants; unit: Participants] | 10 | 10 | 20
Donor Type [Count of Participants; unit: Participants]
  Deceased | 2 | 3 | 5
  Living-unrelated | 2 | 5 | 7
  Living-related | 6 | 2 | 8
Duration of Pre-transplant dialysis [Mean (Standard Deviation); unit: days] | 45.8 (36.6) | 55.8 (46.8) | 50.8 (41.7)
Cause of End Stage Renal Disease [Count of Participants; unit: Participants]
  hypertension (HTN) | 3 | 4 | 7
  diabetes mellitus (DM) | 2 | 0 | 2
  DM + HTN | 4 | 3 | 7
  Other | 1 | 3 | 4
Hospital stay in days [Median (Full Range); unit: days] | 7 [6 to 21] | 6.5 [5 to 17] | 6.75 [5.5 to 19]
Body Mass Index at Transplant [Mean (Standard Deviation); unit: kg/m2] | 38.2 (5.2) | 43.4 (6.8) | 40.8 (6)
Weight at Transplant [Mean (Standard Deviation); unit: kg] | 116.8 (30.2) | 136.4 (30.5) | 126.6 (30.35)
Ideal Body Weight [Mean (Standard Deviation); unit: kg] | 68 (13.3) | 71.5 (11.8) | 69.75 (12.55)
Adjusted Body Weight [Mean (Standard Deviation); unit: kg] | 86.7 (19.5) | 97.5 (17.9) | 92.1 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Tacrolimus Exposure (AUC-0-24)) in Obese Patients Who Received an Initial TAC -ER Dose of 0.15 mg/kg Using aBW Versus IBW
Description: Difference in tacrolimus exposure (area under the concentration-time curve from time 0 to 24 hours (AUC-0-24)) in obese patients who received an initial TAC -ER dose of 0.15 mg/kg using aBW versus IBW
Time Frame: Days 1-14
Population: This study randomized de novo kidney transplant recipients who were at least 18 years of age and obese as evidenced by a BMI ≥ 30 on the day of transplantation.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Ideal Body Weight- Tacrolimus Extended Release | Adjusted Body Weight-Tacrolimus Extended Release
Number analyzed (Participants) | 10 | 10
ng•h/mL
  day 1 AUC 0-24 | 115.2 (51.3) | 90.0 (51.2)
  day 7 AUC 0-24 | 268.3 (59.9) | 269.3 (101.1)
  day 14 AUC 0-24 | 355.0 (75.4) | 267.3 (101.3)
Statistical Analysis 1: Comparison: Ideal Body Weight- Tacrolimus Extended Release vs Adjusted Body Weight-Tacrolimus Extended Release; Test type: Other; p = 0.29, t-test, 2 sided

2. Secondary Outcome: Difference in Time to Therapeutic Level
Description: Difference in the time to a therapeutic tacrolimus trough level in the aBW group compared to the IBW group.
Time Frame: Days 1 to 7
Measure: Mean (Standard Deviation); unit: days
Groups:
- Ideal Body Weight: Astagraf 0.15 mg/kg/day based on ideal body weight (IBW)
- Adjusted Body Weight: Astagraf 0.15 mg/kg/day based on adjusted body weight (aBW)
Arm/Group | Ideal Body Weight | Adjusted Body Weight
Number analyzed (Participants) | 10 | 10
days | 4.9 (3.1) | 5.1 (4.0)
Statistical Analysis 1: Comparison: Ideal Body Weight vs Adjusted Body Weight; Test type: Other; p = 0.90, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year 6 months
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information is the same from clinicaltrials.gov.
Arm/Group | Ideal Body Weight- Tacrolimus Extended Release | Adjusted Body Weight-Tacrolimus Extended Release
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ideal Body Weight- Tacrolimus Extended Release (N=10) | Adjusted Body Weight-Tacrolimus Extended Release (N=10)
Edema (Cardiac disorders) | 2 (2) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Bladder spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tremor (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Delayed graft function (Renal and urinary disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02444143/Prot_SAP_000.pdf